CLINICAL TRIAL: NCT00035724
Title: Monitoring Community Trends in Heart Failure
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1039; R37HL069874 (NIH)
Record Dates: First submitted 2002-05-04; First posted 2002-05-06 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-05

CONDITIONS: Cardiovascular Diseases; Heart Failure, Congestive; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Failure; Heart Diseases

SUMMARY:
To examine temporal trends from 1995 and 2000 in the incidence rates of heart failure, its therapeutic management, and changes over time in the hospital and long-term survival of patients with heart failure.

DETAILED DESCRIPTION:
BACKGROUND:

Heart failure is estimated to contribute to nearly 1 million hospitalizations and approximately 250,000 deaths annually in the U.S. The number of new cases of heart failure in the U.S. is estimated to exceed 400,000 annually. Though reliable estimates of the magnitude, incidence, and mortality of heart failure remain sorely lacking, heart failure is associated with a grim prognosis. However, little recent data exist, particularly from a community-wide perspective, to determine whether the incidence or survival associated with heart failure, and the management of this clinical syndrome, has changed over time.

DESIGN NARRATIVE:

The study uses residents of the Worcester (MA) metropolitan area (1990 census 437,000) and examines changes over time in these and additional outcomes for patients with validated heart failure during 1995 and 2000. Complimenting the hospital surveillance of heart failure, newly diagnosed cases of heart failure occurring in members of the largest HMO in Central Massachusetts during 1995 and 2000 will be identified and monitored over time. To accomplish the study objectives, the medical records of residents of the Worcester metropolitan area hospitalized with a discharge diagnosis of heart failure and related diagnostic rubrics will be individually reviewed and validated according to pre-established diagnostic criteria. The use of traditional criteria for heart failure as well as development of new criteria for the epidemiological study of heart failure will be an important focus of this observational study. Records for additional hospitalizations and death certificates will be reviewed to examine trends in long-term survival of discharged hospital patients through the year 2005.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Goldberg — University of Massachusetts, Worcester

REFERENCES:
- [Background] Goldberg RJ, Spencer FA, Farmer C, Meyer TE, Pezzella S. Incidence and hospital death rates associated with heart failure: a community-wide perspective. Am J Med. 2005 Jul;118(7):728-34. doi: 10.1016/j.amjmed.2005.04.013. PMID 15989906
- [Background] Goldberg RJ, Glatfelter K, Burbank-Schmidt E, Farmer C, Spencer FA, Meyer T. Trends in mortality attributed to heart failure in Worcester, Massachusetts, 1992 to 2001. Am J Cardiol. 2005 Jun 1;95(11):1324-8. doi: 10.1016/j.amjcard.2005.01.076. PMID 15904637